CLINICAL TRIAL: NCT07119788
Title: Investigating the Cognitive, Vascular, and Metabolic Benefits of a Vitamin- and Mineral-Enhanced Haskap Berry Dietary Supplement
Brief Title: Investigating the Effects of a Haskap Berry Supplement on Cognitive Health
Acronym: HACVAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Haskapa Ltd (Unknown)
Responsible Party: Principal Investigator, Prof Claire Williams, Professor, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UREC 25/08; FA2_24-11 (Other Grant/Funding Number: BBSRC OIRC STAR Hub feasibility award)
Record Dates: First submitted 2025-08-05; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Cognition
Keywords: Cognition; Mood; Stress; Vascular; Blood glucose; Haskap berries

STUDY DESIGN:
Intervention Model Description: Participants will be allocated to receive either a vitamin- and mineral-enhanced haskap berry powdered supplement, pure haskap berry powder, or a calorie matched placebo powder
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): 30 participants to receive daily 6g servings of a calorie-matched powder, artificially coloured and flavoured to resemble berry powder
  Interventions: Dietary Supplement: Placebo
- Pure haskap berry powder (Experimental): 30 participants to receive daily 6g servings of a pure, freeze-dried haskap berry powder
  Interventions: Dietary Supplement: Pure haskap berry powder
- Vitamin- and mineral-enhanced haskap berry powder (Experimental): 30 participants to receive daily 6g servings of a vitamin- and mineral-enhanced haskap berry powder (fortified with potassium iodide, zinc bisglycinate, vitamin B5, and vitamin B12
  Interventions: Dietary Supplement: Vitamin-and mineral-enhanced haskap berry powder

INTERVENTIONS:
Dietary Supplement: Placebo — 6g serving of a calorie-matched powder, artificially coloured and flavoured to resemble berry powder
  Arms: Placebo
Dietary Supplement: Pure haskap berry powder — 6g serving of a pure, freeze-dried haskap berry powder
  Arms: Pure haskap berry powder
Dietary Supplement: Vitamin-and mineral-enhanced haskap berry powder — 6g serving of a vitamin- and mineral-enhanced haskap berry powder (fortified with potassium iodide, zinc bisglycinate, vitamin B5, and vitamin B12
  Arms: Vitamin- and mineral-enhanced haskap berry powder

SUMMARY:
This study aims to investigate the postprandial (2h) and longer term (4 week) effects of a haskap berry supplement on cognitive, vascular, and metabolic function in healthy ageing adults aged 50+.

DETAILED DESCRIPTION:
This project aims to investigate the acute benefits (during the immediate post prandial period up to 2 hours) and chronic benefits (following 4 weeks daily supplementation) of a vitamin- and mineral-enhanced haskap berry supplement made from freeze-dried, powdered haskap berries. The main objective of this study is to trial the product in older adults aged 50+ to determine any cognitive, metabolic, or cardiovascular benefits over and above haskap powder alone or a placebo powder. The study will involve a screening visit and two testing visits, 4 weeks apart. For the 24 hours prior to each test visit, participants are asked to follow a low polyphenol diet. They are requested not to consume any food or drinks except water after 8.30pm, and on the morning of test visits to only consume one slice of buttered white toast and a glass of water prior to attending the visit. During the testing visits, cognitive and mood battery tests (to include measures of memory, executive functions, and stress, will be taken at baseline, at 2 hours following the consumption of the supplement as part of a meal, and again at 4 weeks following daily consumption of the supplement added to their usual diet. Blood glucose finger pricks will be recorded at each time point along with FMD (a measure of vascular reactivity).

ELIGIBILITY:
Inclusion Criteria:

* 50+ years old
* Fruit & veg intake less than or equal to 4 servings per day
* Adequate English language and visual & auditory acuity to perform the cognitive tasks
* Normal BMI for age

Exclusion Criteria:

* Being diagnosed with psychological or psychiatric disorders
* ADHD or dyslexia
* Any food allergy or intolerance
* Use of medications and dietary supplements that may impact study results
* Antibiotic use within the last 3 months
* Adherence to vegan or vegetarian diets, or other specific diets that may impact study outcomes
* Conditions altering absorption of nutrients (e.g. celiac disease)
* Being diagnosed with cardiometabolic disease (including type II diabetes and cardiovascular disease), or suffer from untreated hypertension or thrombosis related disorders
* Taking blood thinners

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Delayed recall (Rey Auditory Verbal Learning Task) | Baseline
  The RAVLT is a verbal learning task that presents participants with 15 words (list A) 5 times, giving participants one minute after each presentation to recall as many words as they can from the list. After 5 presentations, a new list (list B) is presented and recalled, and finally participants are asked (without hearing list A again) to recall as many words as they can from list A. After a 30 minute period, participants are asked to think back to the task and recall as many words as possible from list A only, providing a measure of delayed recall.
Delayed recall (Rey Auditory Verbal Learning Task) | 2 hours
  The RAVLT is a verbal learning task that presents participants with 15 words (list A) 5 times, giving participants one minute after each presentation to recall as many words as they can from the list. After 5 presentations, a new list (list B) is presented and recalled, and finally participants are asked (without hearing list A again) to recall as many words as they can from list A. After a 30 minute period, participants are asked to think back to the task and recall as many words as possible from list A only, providing a measure of delayed recall.
Delayed recall (Rey Auditory Verbal Learning Task) | 4 weeks
  The RAVLT is a verbal learning task that presents participants with 15 words (list A) 5 times, giving participants one minute after each presentation to recall as many words as they can from the list. After 5 presentations, a new list (list B) is presented and recalled, and finally participants are asked (without hearing list A again) to recall as many words as they can from list A. After a 30 minute period, participants are asked to think back to the task and recall as many words as possible from list A only, providing a measure of delayed recall.

SECONDARY OUTCOMES:
Rate of learning (Rey Auditory Verbal Learning Task) | Baseline
  The RAVLT is a verbal learning task that presents participants with 15 sequential words (list A) 5 times, giving participants one minute after each presentation to recall as many words as they can from the list. Scores are recorded as a percentage of accuracy, and the rate of learning is determined through change in accuracy across the 5 recalls.
Rate of learning (Rey Auditory Verbal Learning Task) | 2 hours
  The RAVLT is a verbal learning task that presents participants with 15 sequential words (list A) 5 times, giving participants one minute after each presentation to recall as many words as they can from the list. Scores are recorded as a percentage of accuracy, and the rate of learning is determined through change in accuracy across the 5 recalls.
Rate of learning (Rey Auditory Verbal Learning Task) | 4 weeks
  The RAVLT is a verbal learning task that presents participants with 15 sequential words (list A) 5 times, giving participants one minute after each presentation to recall as many words as they can from the list. Scores are recorded as a percentage of accuracy, and the rate of learning is determined through change in accuracy across the 5 recalls.
Word recognition (Rey Auditory Verbal Learning Task) | Baseline
  Following the delayed word recall, words from list A, list B and novel words are displayed sequentially on the screen and participants are asked to indicate which words were from list A only.
Word recognition (Rey Auditory Verbal Learning Task) | 2 hours
  Following the delayed word recall, words from list A, list B and novel words are displayed sequentially on the screen and participants are asked to indicate which words were from list A only.
Word recognition (Rey Auditory Verbal Learning Task) | 4 weeks
  Following the delayed word recall, words from list A, list B and novel words are displayed sequentially on the screen and participants are asked to indicate which words were from list A only.
Modified Attention Network Task (MANT) | Baseline
  This task examines execution function, attention and inhibition. Participants respond to a centrally presented target arrow pointing to the left or the right by pressing the corresponding key on the keyboard. The target arrow is flanked by arrows that point in the same (congruent) or opposite (incongruent) direction. Previous studies have found that participants show larger latencies and more errors on incongruent trials when compared with congruent trials due to the conflicting interference of the incongruently facing arrows. Response latencies to congruent trials reflect processing speed, while errors on incongruent trials indicate susceptibility to interference. In this study participants will be presented with two blocks of the MANT - one normal block, and one block with the addition of serial 3s. In the serial 3s block, participants will be asked to count backwards in 3s out loud while continuing to perform the MANT, increasing the level of cognitive demand.
Modified Attention Network Task (MANT) | 2 hours
  This task examines execution function, attention and inhibition. Participants respond to a centrally presented target arrow pointing to the left or the right by pressing the corresponding key on the keyboard. The target arrow is flanked by arrows that point in the same (congruent) or opposite (incongruent) direction. Previous studies have found that participants show larger latencies and more errors on incongruent trials when compared with congruent trials due to the conflicting interference of the incongruently facing arrows. Response latencies to congruent trials reflect processing speed, while errors on incongruent trials indicate susceptibility to interference. In this study participants will be presented with two blocks of the MANT - one normal block, and one block with the addition of serial 3s. In the serial 3s block, participants will be asked to count backwards in 3s out loud while continuing to perform the MANT, increasing the level of cognitive demand.
Modified Attention Network Task (MANT) | 4 weeks
  This task examines execution function, attention and inhibition. Participants respond to a centrally presented target arrow pointing to the left or the right by pressing the corresponding key on the keyboard. The target arrow is flanked by arrows that point in the same (congruent) or opposite (incongruent) direction. Previous studies have found that participants show larger latencies and more errors on incongruent trials when compared with congruent trials due to the conflicting interference of the incongruently facing arrows. Response latencies to congruent trials reflect processing speed, while errors on incongruent trials indicate susceptibility to interference. In this study participants will be presented with two blocks of the MANT - one normal block, and one block with the addition of serial 3s. In the serial 3s block, participants will be asked to count backwards in 3s out loud while continuing to perform the MANT, increasing the level of cognitive demand.
Task Switching Task | Baseline
  This task requires executive function and sustained attention, and provides a measure of cognitive flexibility. Participants view a circle with 8 equally spaced radii, 2 of which form a bold bisecting line. Numbers are chosen randomly from a set of 1-4 & 6-9 and displayed sequentially in a clockwise direction. A response of higher or lower than 5 is made for trials below the bold line, and even or odd for numbers above the line. Outcome measures include overall accuracy and reaction time (RT) on correct trials, as well as accuracy and RT on trials where there is a 'switch cost' from stimuli moving from below to above the bold line and vice versa.
Task Switching Task | 2 hours
  This task requires executive function and sustained attention, and provides a measure of cognitive flexibility. Participants view a circle with 8 equally spaced radii, 2 of which form a bold bisecting line. Numbers are chosen randomly from a set of 1-4 & 6-9 and displayed sequentially in a clockwise direction. A response of higher or lower than 5 is made for trials below the bold line, and even or odd for numbers above the line. Outcome measures include overall accuracy and reaction time (RT) on correct trials, as well as accuracy and RT on trials where there is a 'switch cost' from stimuli moving from below to above the bold line and vice versa.
Task Switching Task | 4 weeks
  This task requires executive function and sustained attention, and provides a measure of cognitive flexibility. Participants view a circle with 8 equally spaced radii, 2 of which form a bold bisecting line. Numbers are chosen randomly from a set of 1-4 & 6-9 and displayed sequentially in a clockwise direction. A response of higher or lower than 5 is made for trials below the bold line, and even or odd for numbers above the line. Outcome measures include overall accuracy and reaction time (RT) on correct trials, as well as accuracy and RT on trials where there is a 'switch cost' from stimuli moving from below to above the bold line and vice versa.
Corsi Block Tapping Task | Baseline
  A standardised assessment of visuospatial working memory. The task comprises nine identical squares fixed in a random arrangement on a screen. Participants observe sequences of between two and nine blocks, which they then reproduce as accurately as possible by clicking with the mouse. Outcomes include number of correct sequences identified as a percentage of accuracy, and number of correct blocks identified (not necessarily in the correct sequence). Four versions of each sequence length are presented during the task. A novel sequence will be presented on each occasion, the order of which will be counterbalanced across participants.
Corsi Block Tapping Task | 2 hours
  A standardised assessment of visuospatial working memory. The task comprises nine identical squares fixed in a random arrangement on a screen. Participants observe sequences of between two and nine blocks, which they then reproduce as accurately as possible by clicking with the mouse. Outcomes include number of correct sequences identified as a percentage of accuracy, and number of correct blocks identified (not necessarily in the correct sequence). Four versions of each sequence length are presented during the task. A novel sequence will be presented on each occasion, the order of which will be counterbalanced across participants.
Corsi Block Tapping Task | 4 weeks
  A standardised assessment of visuospatial working memory. The task comprises nine identical squares fixed in a random arrangement on a screen. Participants observe sequences of between two and nine blocks, which they then reproduce as accurately as possible by clicking with the mouse. Outcomes include number of correct sequences identified as a percentage of accuracy, and number of correct blocks identified (not necessarily in the correct sequence). Four versions of each sequence length are presented during the task. A novel sequence will be presented on each occasion, the order of which will be counterbalanced across participants.
Flow mediated dilation (FMD) | Baseline
  Participants will complete FMD assessment prior to each cognitive task battery (baseline, 2 hours, 4 weeks). FMD is a non-invasive ultrasound technique that measures how the brachial artery dilates in response to increased blood flow following occlusion. Participants are required to lie down for 15 minutes before scanning commences. The procedure then takes 9 minutes: the brachial artery is first scanned for 1 minute, a blood pressure cuff is then inflated on the forearm for 5 minutes, before being released and the artery scanned for a further 3 minutes. This data will be analysed using Cardiovascular Suit. During FMD, laser doppler flowometry (LDF) will also be measured using the index finger of the right arm and analysed for % PORH (post occlusive reactive hyperaemia), measured in flux units .
Flow mediated dilation (FMD) | 2 hours
  Participants will complete FMD assessment prior to each cognitive task battery (baseline, 2 hours, 4 weeks). FMD is a non-invasive ultrasound technique that measures how the brachial artery dilates in response to increased blood flow following occlusion. Participants are required to lie down for 15 minutes before scanning commences. The procedure then takes 9 minutes: the brachial artery is first scanned for 1 minute, a blood pressure cuff is then inflated on the forearm for 5 minutes, before being released and the artery scanned for a further 3 minutes. This data will be analysed using Cardiovascular Suit. During FMD, laser doppler flowometry (LDF) will also be measured using the index finger of the right arm and analysed for % PORH (post occlusive reactive hyperaemia), measured in flux units .
Flow mediated dilation (FMD) | 4 weeks
  Participants will complete FMD assessment prior to each cognitive task battery (baseline, 2 hours, 4 weeks). FMD is a non-invasive ultrasound technique that measures how the brachial artery dilates in response to increased blood flow following occlusion. Participants are required to lie down for 15 minutes before scanning commences. The procedure then takes 9 minutes: the brachial artery is first scanned for 1 minute, a blood pressure cuff is then inflated on the forearm for 5 minutes, before being released and the artery scanned for a further 3 minutes. This data will be analysed using Cardiovascular Suit. During FMD, laser doppler flowometry (LDF) will also be measured using the index finger of the right arm and analysed for % PORH (post occlusive reactive hyperaemia), measured in flux units .
Blood glucose | Baseline
  Blood glucose will be measured before each cognitive task battery (baseline, 2h, 4 weeks) using finger prick capillary sampling and an Accu-Chek Instant blood glucose monitor.
Blood glucose | 2 hours
  Blood glucose will be measured before each cognitive task battery (baseline, 2h, 4 weeks) using finger prick capillary sampling and an Accu-Chek Instant blood glucose monitor.
Blood glucose | 4 weeks
  Blood glucose will be measured before each cognitive task battery (baseline, 2h, 4 weeks) using finger prick capillary sampling and an Accu-Chek Instant blood glucose monitor.
Blood pressure | Baseline
  Average (triplicate) resting brachial left arm cuffed systolic and diastolic blood pressure mmHg.
Blood pressure | 2 hours
  Average (triplicate) resting brachial left arm cuffed systolic and diastolic blood pressure mmHg.
Blood pressure | 4 weeks
  Average (triplicate) resting brachial left arm cuffed systolic and diastolic blood pressure mmHg.
Positive and Negative Affect Schedule (PANAS-X) performance | Baseline
  A validated self-report measure of affective state. The PANAS comprises of two distinct affective states (positive and negative), as well as 11 individual affective states (fear, guilt, sadness, surprise, hostility, shyness, joviality, self-assurance, attentiveness, fatigue and serenity). Subjects use a Likert scale from 1 - 5 to indicate how the word relates to how they are currently feeling. As this analysis is exploratory all affective states will be explored.
Positive and Negative Affect Schedule (PANAS-X) performance | 2 hours
  A validated self-report measure of affective state. The PANAS comprises of two distinct affective states (positive and negative), as well as 11 individual affective states (fear, guilt, sadness, surprise, hostility, shyness, joviality, self-assurance, attentiveness, fatigue and serenity). Subjects use a Likert scale from 1 - 5 to indicate how the word relates to how they are currently feeling. As this analysis is exploratory all affective states will be explored.
Positive and Negative Affect Schedule (PANAS-X) performance | 4 weeks
  A validated self-report measure of affective state. The PANAS comprises of two distinct affective states (positive and negative), as well as 11 individual affective states (fear, guilt, sadness, surprise, hostility, shyness, joviality, self-assurance, attentiveness, fatigue and serenity). Subjects use a Likert scale from 1 - 5 to indicate how the word relates to how they are currently feeling. As this analysis is exploratory all affective states will be explored.
Stress (Perceived Stress Scale) | Baseline
  Stress scores will be measured using the Perceived Stress Scale (PSS) at baseline and 4 weeks
Stress (Perceived Stress Scale) | 4 weeks
  Stress scores will be measured using the Perceived Stress Scale (PSS) at baseline and 4 weeks

OTHER OUTCOMES:
IQ (Raven's Progressive Matrices) | Baseline
  The Raven's is a non-verbal intelligence test designed to assess abstract reasoning and fluid intelligence which provides a single score (the sum of correct answers). Ravens will be included in the present study at baseline as a measure of IQ, which may later be utilised as a covariate when analysing the cognitive data.
Habitual diet (Epic-Norfolk Food Frequency Questionnaire) | Baseline
  The FFQ is a validated tool for gauging the average habitual dietary intake of micro and macronutrients of an individual in the UK. Data will be processed using the FETA software.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Williams, Principal Investigator — University of Reading
Locations (1):
- Nutrition, Cognition & Health Lab, School of Psychology and Clinical Language Sciences, University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All relevant study outcomes described in the Ethics Review Application Form, including demographics, anthropometrics, cognitive performance, blood glucose, and FMD data, will be preserved and made available via a data repository, such as the University of Reading data repository, in anonymised form, so that they can be consulted and re-used by others.